CLINICAL TRIAL: NCT05050682
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE STUDY TO INVESTIGATE THE MASS BALANCE, METABOLISM AND EXCRETION OF [14C]-PF-07304814 IN HEALTHY PARTICIPANTS USING A 14C-MICROTRACER APPROACH
Brief Title: Study to Investigate the Mass Balance, Metabolism, and Excretion of [14C]-PF-07304814 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4611003; NCT05050682 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: COVID-19; SARS-COV-2; Viral Disease
MeSH Terms: conditions — COVID-19; Virus Diseases | interventions — lufotrelvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-07304814 (Experimental): PF-07304814 is an anti-viral, formulated for intravenous delivery
  Interventions: Drug: PF-07304814

INTERVENTIONS:
Drug: PF-07304814 — PF-07304814 is an anti-viral, formulated for intravenous delivery

SUMMARY:
This open-label, single dose study in approximately 5 healthy male and female (of non childbearing potential only) participants has been designed to characterize mass balance and further the understanding of human pharmacokinetics, metabolism, and excretion of PF 07304814 administered at a dose of 500 mg [14C] PF-07304814 containing approximately 420 nCi [14C] PF-07304814 as a constant-rate, continuous IV infusion over 24 hours

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.
2. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECGs.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. BMI of 18 to 32 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
4. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
5. Participants who have received a COVID-19 vaccine within the past 2 weeks; and/or participants who are scheduled to receive a second COVID-19 vaccination dose during the in-clinical period of this study.
6. A positive urine drug test.
7. Total 14C radioactivity measured in plasma exceeding 11 mBq/mL at "Screening" .
8. Females who are breastfeeding.
9. History of tobacco or nicotine use within 3 months prior to dosing, or a positive cotinine at screening or Day -1.
10. Participants enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry (ie, occupational exposure of 5 rem per year).

13. Participants whose occupation requires exposure to radiation or monitoring of radiation exposure.

14. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Fortrea Clinical Research Unit - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4611003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5 participants were assigned to the study intervention and completed the study.
Groups:
- 14C-PF-07304814 500 mg IV: Participants received 500 mg PF-07304814 containing approximately 420 nCi [14C] PF-07304814 starting at approximately 08:00 hour (±2 hours), administered as a single, 24-hour constant-rate, continuous IV infusion.
Period: Overall Study
Arm/Group | 14C-PF-07304814 500 mg IV
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.40 (10.50)
Age, Continuous [Median (Full Range); unit: years] | 40.0 [23 to 48]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-25 years | 1
  26-35 years | 1
  36-45 years | 2
  >45 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Mean (SD) Amount of [14C] Recovered in Urine, as a Percent of the Total [14C] Dose Administered
Description: This is to confirm mass balance and characterize the routes of elimination of [14C]-PF-07304814 and drug related materials following 420 nCi/500 mg dose of [14C] PF-07304814.
Time Frame: from pre-dose to 216h post the start of infusion
Population: Mass Balance Analysis Set: The mass balance analysis set was defined as all participants who received study intervention and who had evaluable total [14C] concentration (urinary and fecal) data and who had no protocol deviations or AEs (such as diarrhea or severe constipation) that might have affected the mass balance analysis.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
percentage of dose | 25.2 (3.3)

2. Primary Outcome: The Mean (SD) Amount of [14C] Recovered in Feces, as a Percent of the Total [14C] Dose Administered
Description: as for outcome 1
Time Frame: from pre-dose to 216h post the start of infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Groups:
- 14C-PF-07304814 500 mg IV: Participants received 500 mg PF-07304814 containing approximately 420 nCi [14C] PF 07304814 starting at approximately 08:00 hour (±2 hours), administered as a single, 24-hour constant-rate, continuous IV infusion.
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
percentage of dose | 34.0 (4.7)

3. Primary Outcome: The Mean (SD) Percentage of [14C] Relative to the Administered Dose in Excreta (Urine + Feces)
Description: as for outcome 1
Time Frame: from pre-dose to 216h post the start of infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
percentage of dose | 59.2 (3.9)

4. Primary Outcome: Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) for Plasma PF-07304814 and Plasma PF-00835231
Description: Area under the concentration-time profile from time zero to the time of the last quantifiable concentration (Clast), using linear/log trapezoidal method.
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the parameters of primary interest in plasma, urine or feces.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ng*hr/mL
  plasma PF-07304814 | 7322 (23)
  plasma PF-00835231 | 22350 (13)

5. Primary Outcome: Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) for Plasma Total [14C]
Description: as for outcome 4
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ngEq*hr/mL | 468800 (16)

6. Primary Outcome: Area Under the Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) for Plasma PF-00835231
Description: Area under the concentration-time profile from time zero extrapolated to infinite time. AUClast + (Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis (if data permit).
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the parameters of primary interest in plasma, urine or feces. Data could not be estimated for AUCinf for the phosphate prodrug PF-07304814 due to the lack of a well characterized terminal elimination phase. A well characterized terminal phase is defined as one with at least 3 data points can be used for log-linear regression, r2 ≥0.9, and AUCextrap% ≤ 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ng*hr/mL
  plasma PF-07304814: number analyzed (Participants) | 0
  plasma PF-00835231 | 22620 (13)

7. Primary Outcome: AUCinf for Plasma Total [14C]
Description: as for outcome 6
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the parameters of primary interest in plasma, urine or feces. AUCinf values were not reported for the total [14C] due to the lack of a well characterized terminal elimination phase. A well characterized terminal phase is defined as one with at least 3 data points can be used for log-linear regression, r2 ≥0.9, and AUCextrap% ≤ 20%.
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 0

8. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Plasma PF-07304814 and Plasma PF-00835231
Description: Maximum observed plasma concentration. This was observed directly from data.
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ng/mL
  plasma PF-07304814 | 359.8 (24)
  plasma PF-00835231 | 1044 (11)

9. Primary Outcome: Cmax for Plasma Total [14C]
Description: Maximum observed plasma concentration. This was observed directly from data.
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ngEq/mL | 8258 (11)

10. Primary Outcome: Time for Cmax (Tmax) for Plasma PF-07304814 and Plasma PF-00835231
Description: Time for Cmax. This was observed directly from data as time of first occurrence.
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
hour
  plasma PF-07304814 | 12 [2.02 to 24.0]
  plasma PF-00835231 | 24.0 [24.0 to 24.0]

11. Primary Outcome: Tmax for Plasma Total 14C
Description: Time for Cmax. This was observed directly from data as time of first occurrence.
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
hour | 24.0 [24.0 to 24.0]

12. Primary Outcome: Obsereved Plasma Concentration at 24 Hours (C24) for Plasma PF-07304814 and Plasma PF-00835231
Description: Obsereved plasma concentration at 24 hours. This was observed directly from data.
Time Frame: 24 hours post the start of infusion
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ng/mL
  plasma PF-07304814 | 313.9 (19)
  plasma PF-00835231 | 1044 (11)

13. Primary Outcome: C24 for Plasma Total [14C]
Description: Obsereved plasma concentration at 24 hours. This was observed directly from data.
Time Frame: 24hours post the start of infusion
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
ngEq/mL | 8258 (11)

14. Primary Outcome: Systematic Clearance (CL) for Plasma PF-07304814
Description: Systemic clearance. This was determined by Dose/AUCinf (if data permit).
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the parameters of primary interest in plasma, urine or feces. CL values were not reported for the phosphate prodrug PF-07304814 due to the lack of a well characterized terminal elimination phase. A well characterized terminal phase is defined as one with at least 3 data points can be used for log-linear regression, r2 ≥0.9, and AUCextrap% ≤ 20%.
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 0

15. Primary Outcome: Steady-state Volume of Distribution Following Intravenous Infusion (Vss) for Plasma PF-07304814
Description: Steady-state volume of distribution following intravenous infusion. This was determined by Vss=CL × [MRT-(infusion time/2)] where MRT is the Mean Residence Time and is calculated as AUMCinf (the area under the first moment curve from time 0 extrapolated to infinite time)/AUCinf (area under the concentration-time profile from time 0 extrapolated to infinite time), if data permit.
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the parameters of primary interest in plasma, urine or feces. Vss values were not reported for the phosphate prodrug PF-07304814 due to the lack of a well characterized terminal elimination phase. A well characterized terminal phase is defined as one with at least 3 data points can be used for log-linear regression, r2 ≥0.9, and AUCextrap% ≤ 20%.
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 0

16. Primary Outcome: Terminal Elimination Half-life (t½) for Plasma PF-00835231
Description: Terminal elimination half-life. This was determined by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve (if data permit).
Time Frame: 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the parameters of primary interest in plasma, urine or feces. Data could not be estimated for t½ for the phosphate prodrug PF-07304814 due to the lack of a well characterized terminal elimination phase. A well characterized terminal phase is defined as one with at least 3 data points can be used for log-linear regression, r2 ≥0.9, and AUCextrap% ≤ 20%.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
hour
  plasma PF-07304814: number analyzed (Participants) | 0
  plasma PF-00835231 | 1.496 (0.30088)

17. Primary Outcome: t½ for Plasma Total [14C]
Description: as for outcome 16
Time Frame: pre-dose, 0.5h, 1h, 2h, 6h, 12h, 24h, 25h, 27h, 32h, 48h, 72h, 96h, 120h, 144h, 216h post the start of infusion
Population: The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the parameters of primary interest in plasma, urine or feces. t½ values were not reported for the total [14C] due to the lack of a well characterized terminal elimination phase.
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 0

18. Secondary Outcome: Percentage of Total Radioactivity in Each Matrix (Plasma, Urine and Feces) of Metabolites of PF-07304814
Description: The percentage of radioactivity collected over the time frame for each metabolite was determined and reported as percentage of total radioactivity in each matrix (plasma, urine and feces).
Time Frame: Predose to maximum of Day 10
Population: The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the parameters of primary interest in plasma, urine or feces. Data reported with measure type "Number" as the values reported represent the measured value from a pooled sample from all participants in the study.
Measure: Number; unit: Percentage of Radioactivity
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Percentage of Radioactivity
  M12: plasma | 0.4
  M8: plasma | 1.1
  M7: plasma | 21.5
  PF-07304814 and epimer: plasma | 21.5
  M6: plasma | 0.4
  PF-00835231: plasma | 9.8
  Epimer (PF-03626560): plasma | 1.3
  m/z 467: urine | 0.3
  M12: urine | 1.7
  M8: urine | 2.3
  M7 (PF-07305457): urine | 5.4
  M11a: urine | 2.1
  M11b: urine | 0.4
  M11c: urine | 0.5
  M11d: urine | 0.6
  M6: urine | 0.3
  m/z 475: urine | 0.3
  PF-00835231: urine | 7.4
  Epimer (PF-03626560): urine | 0.6
  m/z 287: urine | 0.4
  Unknown: feces | 0.4
  m/z 491: feces | 0.4
  m/z 487: feces | 0.4
  M1 (PF-07307659): feces | 0.8
  M6: feces | 2.6
  m/z 475: feces | 0.2
  PF-00835231: feces | 0.4
  Epimer (PF-03626560): feces | 0.9

19. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-Emergent Adverse Event if the event started during the effective duration of treatment. All events that start on or after the first dosing day and time/ start time, if collected, but before the last dose plus the lag time (28 days) will be flagged as TEAEs. A serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent or significant disability/incapacity, 5. was a congenital anomaly/birth defect, 6. was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, is considered serious, and other situations defined in the protocol
Time Frame: From first dose up to 28-35 days from administration of the dose of study intervention (maximum of 35 days)
Population: The safety analysis set includes all participants assigned to study intervention and who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Participants
  all causality AEs | 3
  treatment related AEs | 2
  serious adverse events | 0

20. Secondary Outcome: Number of Subjects With Vital Signs Data Meeting Categorical Summarization Criteria
Description: The following abnormality criteria were applied: diastolic blood pressure: value < 50 mmHg, change >=20 mmHg increase/decrease; systolic blood pressure: value < 90 mmHg, change >= 30 mmHg increase/decrease; pulse rate: value< 40 beats per minute, value > 120 beats per minute.
Time Frame: from Screening (Day-42 to Day-2) to 216h or early termination/discontinuation
Population: All participants assigned to study intervention and who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Participants | 0

21. Secondary Outcome: Number of Subjects With Laboratory Test Abnormalities (Without Regards to Baseline Abnormality)
Description: Safety laboratory assessments including urinalysis, hematology, and chemistry were performed at the indicated time-points. All the safety laboratory samples must be collected following at least a 4 hour fast.
Time Frame: From Screening (Day-42 to Day-2) to 216h or early termination/discontinuation
Population: All participants assigned to study intervention and who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Participants | 1

22. Secondary Outcome: Number of Subjects With Electrocardiogram (ECG) Data Meeting Categorical Summarization Criteria
Description: ECG endpoints meeting the criteria of potential clinical concern were summarized by treatment using categories as defined:PR interval (msec): value >280, %change >= 25%, %change >= 50%; QRS complex (msec): value > 120; QT interval (msec): value > 500; QTcF (msec): 450 < value <=480, 480 <value <= 500, 30 <= increase <= 60, increase >60.
Time Frame: From Screening (Day-42 to Day-2) to 216h or early termination/discontinuation
Population: All participants assigned to study intervention and who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 14C-PF-07304814 500 mg IV
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: From the first dose to 28-35 days from administration of the dose of study intervention (maximum of 35 days)
Description: Participants were only counted once per treatment for each category.
Arm/Group | 14C-PF-07304814 500 mg IV
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14C-PF-07304814 500 mg IV (N=5)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT05050682/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05050682/SAP_001.pdf